CLINICAL TRIAL: NCT00004660
Title: Phase II Randomized Controlled Study of Sequential Orbital Radiotherapy for Graves' Ophthalmopathy
Brief Title: Randomized Study of Sequential Orbital Radiotherapy for Graves' Ophthalmopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 199/11860; MAYOC-1889200 (Other: Mayo Clinic); R01DK042822 (NIH)
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Graves' Disease
Keywords: Graves' disease; thyroid disease; endocrine disorders; rare disease
MeSH Terms: conditions — Graves Disease; Thyroid Diseases; Endocrine System Diseases; Rare Diseases | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy (Experimental)
  Interventions: Radiation: Radiotherapy
- Sham treatment (Sham Comparator)
  Interventions: Radiation: Sham treatment

INTERVENTIONS:
Radiation: Radiotherapy
  Arms: Radiotherapy
Radiation: Sham treatment
  Arms: Sham treatment

SUMMARY:
OBJECTIVES: I. Evaluate the effects of 20 Gy of external-beam radiotherapy to 1 orbit vs. the untreated orbit at 3 and 6 months after therapy in patients with Graves' ophthalmopathy.

II. Evaluate whether 20 Gy of external-beam radiotherapy delivered to the second orbit 6 months later in the course of the disease produces effects of equal magnitude to those observed when the first orbit was treated.

III. Relate the magnitude of treatment effects to the time since onset of eye symptoms.

IV. Evaluate whether characteristics of radiation retinopathy are present 3 years after orbital radiotherapy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: The posterior region of 1 orbit is irradiated over 2 weeks with supervoltage equipment. The other orbit is treated 6 months later. The sequence of therapy is randomly assigned.

The untreated eye receives a simultaneous sham treatment during each radiotherapy session.

Patients are followed at 3, 6, 9, 12, and 36 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Firm diagnosis of Graves' disease with normal thyroid function, i.e.: Thyroid-stimulating immunoglobulin positive Thyroxine 5-12.5 micrograms/dL Tri-iodothyronine 80-180 nanograms/dL Thyroid-stimulating hormone 0.2-8 milli-International unit (mIU/L) Euthyroid due to therapy acceptable Ophthalmopathy meeting at least 3 of the following criteria: Chemosis or lid edema Lid lag, lid retraction, or restrictive lagophthalmos Proptosis at least 20 mm by Krahn exophthalmometry in at least 1 eye Less than 4 mm discrepancy between eyes Patient perception of "stare" or "bulge" Extraocular muscle motion restriction in 1 or both eyes on clinical exam or by patient report of diplopia at extremes of gaze Extraocular muscle enlargement on computerized tomography (previous study results acceptable) Mild to moderate ophthalmopathy, i.e.: Orbital pain Lacrimation Photophobia Visual blurring or diplopia No optic neuropathy, i.e.: Afferent pupillary defect Impaired color vision on D-15 testing (unless congenital color perception deficiency) Visual field defect Impaired visual acuity No corneal ulcers --Prior/Concurrent Therapy-- No prior external-beam radiotherapy to the head and neck At least 2 weeks since corticosteroids --Patient Characteristics-- No prior head and neck tumors No diabetes No pregnant women

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 1993-06; Primary Completion 1998-01 (Actual); Study Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
Orbital Volume | 1 year
  Orbital fat and muscle volumes

CONTACTS AND LOCATIONS:
Overall Officials: Colum A. Gorman, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Gorman CA, Garrity JA, Fatourechi V, Bahn RS, Petersen IA, Stafford SL, Earle JD, Forbes GS, Kline RW, Bergstralh EJ, Offord KP, Rademacher DM, Stanley NM, Bartley GB. A prospective, randomized, double-blind, placebo-controlled study of orbital radiotherapy for Graves' ophthalmopathy. Ophthalmology. 2001 Sep;108(9):1523-34. doi: 10.1016/s0161-6420(01)00632-7. PMID 11535445